CLINICAL TRIAL: NCT06782204
Title: Variability of Sulfotransferase Activity in Humans: an Approach to Improve Predictive Drug Response Part II: Analysis of Interindividual Variation in Hypertensive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital da Luz, Portugal (Other)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HL_001_2019 v1
Record Dates: First submitted 2020-07-01; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2020-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): At visit 2, complying subjects will receive a tablet containing 1 gram of paracetamol and have blood and urine samples collected 2 hours after administration.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — At visit 2, complying subjects will receive a tablet containing 1 gram of paracetamol and have blood and urine samples collected 2 hours after administration.

SUMMARY:
An open-label, single center, nonrandomized clinical study in hypertensive patients, with intervention, over a 5-week period. After written informed consent, subjects will undergo screening evaluations, including blood and urine sampling (Visit 1). After visit 1, subjects who meet the selection criteria will enter a run-in period where they will receive paracetamol 1g tablet and collect blood and urine samples 2 hours afterwards (visit 2). A final visit for safety assessment will take place at week 5 (visit 3).

Blood and urine samples will be used to quantify paracetamol and its metabolites.

DETAILED DESCRIPTION:
Current approaches to the personalization of hypertension treatment focus primarily on genome sequences and several recent studies have provided insights into the genetic regulation of hypertension. Genome sequences alone, however, do not account for environmental and lifestyle factors that also contribute to hypertension and other common and complex cardiovascular and renal diseases. (Kotchen et al. 2016) The field of hypertension needs clinically applicable phenotyping methods permitting inferences about pathophysiology and expected treatment response.

SULT are at the crossroad of metabolic pathways of catecholamines, drugs including antihypertensives and diverse environmental xenobiotics. Furthermore, SULT display wide interindividual variability, accounted for by ethnically distributed genetic variation (SNPs and CNV), regulation by nuclear receptors, PAPS availability and inhibition by various drugs and environmental compounds.(Marto et al. 2017) We hypothesize that sulfonation varies between hypertensive subjects and low sulfonation phenotypes could be related to deficient inactivation of catecholamines, influencing the pathophysiology of hypertension. We also anticipate that the sulfonation phenotype of an individual could determine response to certain antihypertensive drugs, whether because they are substrates of SULT, inhibitors of SULT or because they interfere with catecholamine activity (adrenergic blockers).

In our current study, we will study the interindividual variation of sulfoconjugation in patients with hypertension. We will quantify SULT activity using the index of sulfonation we previously described (Marto et al. unpublished), built with the mass spectrometry urinary metabolites of paracetamol, our probe substrate. We will look for associations between patients' characteristics and sulfonation phenotype and for differences in SULT activity in subgroups of patients, defined according to concurrent comorbidities and therapeutic regimen.

We expect to find individuals at the extremes of sulfonation phenotype (high and low sulfonators), with low sulfonators having more severe forms of hypertension, requiring a higher number of antihypertensive drugs.(Williams et al. 2018) If confirmed, management of hypertension in this subpopulation of patients could include induction of SULT activity or avoidal of SULT inhibitors.

Accordingly, our purpose is to explore the clinical significance of the variation of SULT activity in hypertensive patients, as an emergent blood pressure and drug response determinant.

This is an exploratory, open-label, nonrandomized clinical trial, spanning over a 6-month period, to assess interindividual variation of SULT activity in patients with arterial hypertension. Subjects must be consenting adults with a diagnosis of arterial hypertension, who comply with the inclusion and exclusion criteria listed below. Patients will be screened at visit 1, and if they meet the inclusion/exclusion criteria they will receive the intervention at visit 2. Baseline blood and urine samples will be collected.

At visit 2, complying subjects will receive a tablet containing 1 gram of paracetamol and have blood and urine samples collected 2 hours after administration. The subjects will come for 3 visits during the study. Visits 1 and 2 must occur from within 0 to 7 days of each other and visit 3 will be scheduled four weeks (± 3 days) after visit 2.

Study visits 1 and 2 will take place at Hospital da Luz in Lisbon, Portugal, and study visit 3 will follow through telephone contact.

The study population will include adult patients with arterial hypertension who will be recruited from the Internal Medicine inpatient and outpatient clinic at Hospital da Luz. Recruitment will continue until 73 patients are included.

Paracetamol and its metabolites will be quantified in plasma and urine samples using liquid chromatography mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the nature of the study and giving written informed consent before any study assessment is performed,
* Able to understand and communicate effectively with study personnel,
* Male or non-pregnant, non-lactating female patients over 18 years of age,
* A diagnosis of hypertension defined either as:

  1. Use of antihypertensive drug(s) and stable dose for at least 2 weeks prior to inclusion,
  2. In untreated patients: office systolic blood pressure values >= 140 mmHg and/ or diastolic blood pressure values >= 90 mmHg,(Williams et al. 2018)
* Have no contraindication for 1 g of oral paracetamol.

Exclusion Criteria:

* Hypersensitivity or idiosyncratic reaction to paracetamol,
* Paracetamol intake in the last seven days before Visit 2,
* Non-steroidal antiinflammatory drug intake,
* Pregnancy or breastfeeding,
* BMI <18 kg/m2,
* History of clinically significant liver disease or liver injury as indicated by abnormal liver enzymes such as ALT, GGT or serum bilirubin (any single parameter may not exceed 2x upper limit of normal),
* Current severe progressive or uncontrolled disease which in the judgement of the investigator renders the patient unsuitable for the study,
* Hospital da Luz employees, NMS|FCM employees, medical students at NMS|FCM and workers or others with a direct dependency on the PI or the sponsor,
* Participation in a clinical study of any investigational product 1 month prior to visit 1 or during the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 6 months
  Coefficient of variation of paracetamol sulfonation index (PSI), a ratio between the measured plasma concentrations of paracetamol sulfate (PS) and PS+ paracetamol glucoronide (PG) + paracetamol (P)

SECONDARY OUTCOMES:
Secondary Outcome Measures | 6 months
  Relationship between PSI and subject characteristics (gender, age, BMI, smoking status, caffeine consumption, alcohol consumption, oral contraceptive use) Differences in PSI between groups of patients with specific comorbidities (diabetes mellitus type 2, obstructive sleep apnea, heart failure, atrial fibrillation) Differences in PSI between groups of patients on defined antihypertensive drug regimens (beta-blocker-based regimen and renin-angiotensin-aldosterone system inhibitors-based regimen) Influence of furosemide treatment on PSI

CONTACTS AND LOCATIONS:
Overall Officials: Natália Marto, MD, Principal Investigator — Hospital da Luz
Locations (1):
- Hospital da Luz, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No